CLINICAL TRIAL: NCT05890924
Title: (WAST-VTE) Intimate Partner Violence as a Risk Factor for Venous Thromboembolism in Women on Combined Oral Contraceptives: a Matched Case-control Study
Brief Title: Intimate Partner Violence as a Risk Factor for Venous Thromboembolism in Women
Acronym: WAST-VTE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2023/JCG-01
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-09

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: First venous thromboembolic event associated with combined oral contraceptives intake
  Interventions: Other: WAST questionnaire
- Controls: regular follow-up of their combined oral contraception
  Interventions: Other: WAST questionnaire

INTERVENTIONS:
Other: WAST questionnaire — WAST questionnaire, designed and validated as a screening tool for violence against women and intimate partner violence.
  (ref: Brown JB, Lent B, Brett PJ, Sas G, Pederson LL. Development of the Woman Abuse Screening Tool for use in family practice. Fam Med. 1996 Jun;28(6):422-8.)

SUMMARY:
The frequency of violence against women, or intimate partner violence (IPV) is more and more underlined and recognized as a cofactor favoring certain somatic and psychic pathologies. However, its incidence in patients with venous thromboembolism (VTE) is unknown and its status as a risk factor is still elusive and ambiguous.

Investigators therefore conducted a matched case-control study consisting of women taking combined oral contraceptives (COC) who were investigated and followed up between 2010 and 2020.

The cases are the patients investigated for their first venous thromboembolic event, The controls were women free of thrombosis who had regular gynecological checkups. Case-control pairs were matched on region of residence, age (+/- 2 years), duration of COC intake (+/- 4 months), COC type (2nd, 3rd or 4th generation).

ELIGIBILITY:
* Patients: first venous thromboembolic event associated with the intake of combined oral contraceptives
* Controls: regular follow-up of their combined oral contraception
* Patient-Control pairs matched on region of residence, age, duration of COC intake, type of COC.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women managed and followed by their respective departments dedicated to the evaluation of the vascular risk in women (Gynecology-Obstetrics + Haematology)
Sampling Method: Non-Probability Sample
Enrollment: 997 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Woman Abuse Screening Tool (WAST) | inclusion
  Self-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe GRIS, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémea, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vandevelde A, Gris JC, Moore GW, Musial J, Zuily S, Wahl D, Devreese KMJ. Added value of antiphosphatidylserine/prothrombin antibodies in the workup of obstetric antiphospholipid syndrome: communication from the ISTH SSC Subcommittee on Lupus Anticoagulant/Antiphospholipid Antibodies. J Thromb Haemost. 2023 Jul;21(7):1981-1994. doi: 10.1016/j.jtha.2023.04.001. Epub 2023 Apr 13. PMID 37061133